CLINICAL TRIAL: NCT00340808
Title: Integration of an Epidemiologic Questionnaire Into Gynecologic Oncology Group Trials: First Project, Protocol 210
Brief Title: Molecular Staging of Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904144; 04-C-N144; NCT00556556 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Epidemiology; Questionnaire; Etiology; Biomarkers
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endometrial cancer cases: endometrial cancer cases

SUMMARY:
This study, sponsored by NCI and the Gynecologic Oncology Group (GOG), will collect tissue samples from women with cancer of the endometrium (lining of the uterus). Researchers will use the samples to learn more about endometrial cancer and develop new treatments and methods of prevention.

Women with endometrial cancer who are suitable candidates for surgery and who have not had prior retroperitoneal surgery or pelvic or abdominal radiation therapy may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood tests, and endometrial biopsy (surgical removal of a small tissue sample) or dilation and curettage (D & C).

Participants will undergo hysterectomy (surgery to remove the uterus) along with removal of both fallopian tubes and ovaries. This is the standard surgical treatment for endometrial cancer. Lymph nodes in the pelvis near the main blood vessel in the abdomen are also removed to determine if the disease has spread to these nodes. If cancer is found involving other sites, the cancer in those areas may also be removed; examination of the tissues will determine if further therapy beyond surgery is needed.

Before surgery, patients will complete a 20-minute questionnaire that includes questions about their background, reproductive history, menstruation and menopause, certain surgeries, birth control pills and hormone replacement therapy, other drugs and medicines, weight and height, smoking, medical history, and family history of cancer.

Some of the tissue removed during surgery, plus a urine sample collected from a catheter bag during surgery, and blood drawn before surgery and at follow-up visits 6 weeks and 3 years after surgery, will be sent to the GOG Tissue Bank in Columbus, Ohio. This bank stores, processes, and distributes biological specimens from patients that agree to participate in studies conducted by the GOG.

Patients will have follow-up visits 6 weeks after surgery, then every 6 months for the next 2 years, followed annually for the next 7 years, for a total 10-year follow-up. The visits will include an examination and questions about health status and treatments received between visits. Patients whose cancer returns or worsens will undergo another tumor biopsy, if possible, at that time.

DETAILED DESCRIPTION:
GOG-210 is a molecular and surgico-pathological staging study of endometrial carcinoma. The overall goal of this pilot protocol is to improve outcome and/or quality of life for patients with endometrial cancer. This fundamental goal will be accomplished through the development of more accurate models of risk, identification of candidate targets for therapeutic intervention and utilization of individualized treatments based on molecular characteristics identified in tumor tissue, normal tissue and/or in readily accessible biological fluids, like serum and urine. This molecular and surgico-pathological staging study is structured to collect tissue, urine, serum, and epidemiologic and clinical data from approximately 3,500 patients with endometrial cancer identified at participating GOG institutions. All of the patients will be surgically-pathologically staged, consistently evaluated, further treated as needed, and followed for up to 10 years after surgery to document further treatment and outcome. A series of independent and integrated research projects will be undertaken to utilize high-throughput methodologies (e.g., genomics and proteomics) and more traditional techniques (e.g., immunoassays) to examine cellular and extracellular factors, including chromosomes, DNA, RNA, proteins, lipids and carbohydrates. The results obtained from the comprehensive laboratory testing performed on these clinical specimens with the clinical and epidemiologic data collected for each GOG-0210 patient will represent an enduring resource for endometrial cancer research to study the factors that control the growth and spread of endometrial cancer, and how to predict response to therapy and risk of disease spread, recurrence and overall survival for patients with this disease. This will be the first implementation of the NCI-developed epidemiologic questionnaire, which will allow GOG protocols to systematically and uniformly collect demographic and epidemiologic data that will enhance the analytic capabilities of this study. If successful, this study will serve as a model for other protocol to implement the same epidemiologic questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with endometrial carcinoma diagnosed by an endometrial biopsy or dilation and curettage who will undergo full surgical staging; all stages, grades and histologic subtypes will be eligible.
* Patients must be suitable candidates for surgery. Patients may also be entered on GOG-2222 (LAP2).
* Patients who have signed an approved Informed Consent.
* Patients who have met the pre-entry requirements specified in the Study Parameters.
* Patients with a prior malignancy (at least 5 years since diagnosis) with no current evidence of disease.

EXCLUSION CRITERIA:

* Patients not considered suitable candidates for surgery.
* Patients who have had prior retroperitoneal surgery.
* Patients who have received prior pelvic or abdominal radiation therapy.
* Patients who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This molecular and surgico-pathological staging study was structured to collect tissue, urine, serum, and epidemiologic and clinical data from approximately 3,500 patients with endometrial cancer identified at participating GOG institutions. All of the patients were surgically-pathologically staged, consistently evaluated, further treated as needed, and will be followed for up to 10 years after surgery to document further treatment and outcome.
Sampling Method: Non-Probability Sample
Enrollment: 5492 (Actual)
Dates: Start 2004-03-19 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
Breast, colorectal, endometrial, and ovarian cancers | Baseline 1992-1993 with 10 years of follow-up (1992-2003)

CONTACTS AND LOCATIONS:
Overall Officials: Britton L Trabert, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Oklahoma, Norman, Oklahoma, United States

REFERENCES:
- [Derived] Hagemann IS, Deng W, Zaino RJ, Powell MA, Gunderson C, Cosgrove C, Mathews C, Pearl ML, Waggoner S, Ghebre R, Lele S, Guntupalli S, Secord AA, Ioffe O, Park K, Rasty G, Singh M, Soslow R, Creasman W, Mutch DG. The presence of an endometrioid component does not alter the clinicopathologic profile or survival of patients with uterine serous cancer: A gynecologic oncology group (GOG/NRG) study of 934 women. Gynecol Oncol. 2021 Mar;160(3):660-668. doi: 10.1016/j.ygyno.2020.12.040. Epub 2021 Jan 8. PMID 33423806
- [Derived] Krill L, Deng W, Eskander R, Mutch D, Zweizig S, Hoang B, Ioffe O, Randall L, Lankes H, Miller DS, Birrer M. Overexpression of enhance of Zeste homolog 2 (EZH2) in endometrial carcinoma: An NRG Oncology/Gynecologic Oncology Group Study. Gynecol Oncol. 2020 Feb;156(2):423-429. doi: 10.1016/j.ygyno.2019.12.003. Epub 2019 Dec 13. PMID 31843273
- [Derived] McMeekin DS, Tritchler DL, Cohn DE, Mutch DG, Lankes HA, Geller MA, Powell MA, Backes FJ, Landrum LM, Zaino R, Broaddus RD, Ramirez N, Gao F, Ali S, Darcy KM, Pearl ML, DiSilvestro PA, Lele SB, Goodfellow PJ. Clinicopathologic Significance of Mismatch Repair Defects in Endometrial Cancer: An NRG Oncology/Gynecologic Oncology Group Study. J Clin Oncol. 2016 Sep 1;34(25):3062-8. doi: 10.1200/JCO.2016.67.8722. Epub 2016 Jun 20. PMID 27325856
- [Derived] Goodfellow PJ, Billingsley CC, Lankes HA, Ali S, Cohn DE, Broaddus RJ, Ramirez N, Pritchard CC, Hampel H, Chassen AS, Simmons LV, Schmidt AP, Gao F, Brinton LA, Backes F, Landrum LM, Geller MA, DiSilvestro PA, Pearl ML, Lele SB, Powell MA, Zaino RJ, Mutch D. Combined Microsatellite Instability, MLH1 Methylation Analysis, and Immunohistochemistry for Lynch Syndrome Screening in Endometrial Cancers From GOG210: An NRG Oncology and Gynecologic Oncology Group Study. J Clin Oncol. 2015 Dec 20;33(36):4301-8. doi: 10.1200/JCO.2015.63.9518. Epub 2015 Nov 9. PMID 26552419
- [Derived] Felix AS, Scott McMeekin D, Mutch D, Walker JL, Creasman WT, Cohn DE, Ali S, Moore RG, Downs LS, Ioffe OB, Park KJ, Sherman ME, Brinton LA. Associations between etiologic factors and mortality after endometrial cancer diagnosis: the NRG Oncology/Gynecologic Oncology Group 210 trial. Gynecol Oncol. 2015 Oct;139(1):70-6. doi: 10.1016/j.ygyno.2015.08.022. Epub 2015 Sep 1. PMID 26341710